CLINICAL TRIAL: NCT04728425
Title: Efficacy and Safety of Subcutaneous Immunoglobulin in Patients With Myasthenia Gravis
Brief Title: Subcutaneous Immunoglobulin for Myasthenia Gravis
Acronym: MG_SCIG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Hans Katzberg, Neurologist, Principle Investigator, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-5378.2
Record Dates: First submitted 2020-07-14; First posted 2021-01-28 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Myasthenia Gravis
Keywords: myasthenia gravis; IVIG; SCIG; subcutaneous immunoglobulin; intravenous immunoglobulin; MG; neuromuscular junction
MeSH Terms: conditions — Myasthenia Gravis | interventions — Hizentra; Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IVIG + SCIG (Active Comparator): This group of MG patients will start with 2g/kg of IVIG on month 1, 1 g/kg of IVIG 4 and then 8 weeks later, and within 2 weeks switch to SCIG treatment
  Interventions: Drug: intravenous immunoglobulin + subcutaneous immunoglobulin (SCIG)
- SCIG alone (Active Comparator): This group of MG patients will start with SCIG alone
  Interventions: Drug: subcutaneous immunoglobulin (SCIG)

INTERVENTIONS:
Drug: subcutaneous immunoglobulin (SCIG) — 20% subcutaneous immunoglobulin
  Other Names: Cuvitru
  Arms: SCIG alone
Drug: intravenous immunoglobulin + subcutaneous immunoglobulin (SCIG) — 10% intravenous immunoglobulin + 20% subcutaneous immunoglobulin
  Other Names: Gammanorm + Cuvitru
  Arms: IVIG + SCIG

SUMMARY:
This is a prospective open-label, randomized, parallel arm clinical trial.

The primary objective of the study is to evaluate the safety and efficacy of Cuvitru 20% subcutaneous immunoglobulin in patients with myasthenia gravis (MG). The secondary objective is to evaluate patient preferences and effects on quality of life when treating MG patients with SCIG. Exploratory objectives are to compare de novo administration starting SCIG directly with those starting with a loading dose of IVIG followed by SCIG administration.

Patients over age 18 with moderate to severe MG with MGFA Class II-IV without contraindications to immunoglobulin will be considered for the study.

All patients will be eligible to enter either arm of the study, Arm 1: 10% Gammagard IVIG followed by 20% Cuvitry SCIG and Arm 2: Cuvitru 20% SCIG alone.

DETAILED DESCRIPTION:
Myasthenia gravis (MG) is an autoimmune neuromuscular condition which can cause fatigable weakness of skeletal muscles including bulbar, ocular, limb, axial and respiratory muscles. Symptoms range from mild, transient double vision and ptosis to severe, life threatening diffuse weakness, and treatments which are immunosuppressive or immunomodulatory have been shown to improve outcome in MG. This includes 10% intravenous immunoglobulin (IVIG), which has previous been shown by our group to improve strength at 2 and 4 weeks in patients with MG. Due to delay in the onset of many immunosuppressives and potential side effects from steroids and other immunosuppressive medications, IVIG is also used in clinical practice as bridging of maintenance therapy until other therapies take effect or the patient stabilizes. In addition, there have been other studies suggesting that 20% subcutaneous immunoglobuin (SCIG) can be helpful to improve strength in patients with MG over a relatively short period of time (6 weeks). Some of these studies are ongoing and are further evaluating the ability of IVIG and SCIG to stabilize or improve strength IVIG in patients with MG, however, there is no current published study evaluating different administration routes of immunoglobulin (IVIG and SCIG) in patients with MG over a longer 6 month follow-up period.

The current study aims to be the first to evaluate 20% Cuvitru SCIG formulation in patients with neuromuscular conditions including MG. The study aim is to evaluate the safety and efficacy of 6 months of 20% SCIG Cuvitru treatment vs three months of 10% IVIG "pre-treatment" followed by 3 months of 20% SCIG Cuvitru treatment. The study will also be the first to use the myasthenia gravis impairment index (MGII) as primary outcome in conjunction with standard MG outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over age 18
2. Patients with a confirmed diagnosis of myasthenia gravis based on clinical criteria including fatiguable weakness and supported by either serological (acetylcholine receptor, muscle specific kinase or anti-low-density lipoprotein receptor- related protein 4 antibodies or electrophysiological testing (repetitive nerve stimulation of single fiber electromyography)
3. Myasthenia Gravis Federation of America class II-IV
4. Moderate to severe myasthenia gravis as defined by a quantitative myasthenia gravis score >10 or generalized myasthenia gravis impairment index score > 11
5. Patient able to give consent and is able and willing to complete all study procedures and activities

Exclusion Criteria:

1. Patients who are pregnant or breastfeeding
2. Patients not able to complete the study procedures or with an alternate diagnosis
3. Patients with recent thymectomy in the past 6 months
4. Patients receiving another biologic agent such as rituximab, belimubab, cyclophosphamide and eculizumab in the past 6 months prior to study entry
5. No IVIG or subcutaneous immunoglobulin within the past month
6. Patients on prednisone who have had alterations in prednisone dose over the past month prior to study entry
7. Patients will previous known allergy or severe adverse reaction to intravenous or subcutaneous immunoglobulin
8. Evidence of renal insufficiency (Cr>1.5 x elevated) or liver disease (transaminases > 2.5 x elevation) at screening.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Myasthenia Gravis Impairment Index Efficacy Outcome | 6 months
  Change in the Myasthenia Gravis Impairment Index (score 0-84, with 84 being the maximal score indicating the most severe MG status) at baseline compared to end of study

SECONDARY OUTCOMES:
Quantitative Myasthenia Gravis Score Efficacy Outcome | 6 months
  Change in the Quantitative Myasthenia Gravis Score (score 0-39, with 39 indicating the most severe clinical findings related to MG) at baseline compared to end of study
Myasthenia Gravis Activities of Daily Living Efficacy Outcome | 6 months
  Change in the MG Activities of Daily Living (score 0-24, with 24 indicating the most severe clinical findings related to MG) at baseline compared to end of study
Myasthenia Gravis Composite Efficacy Outcome | 6 months
  Change in the Myasthenia Gravis Composite Score (score 0-50, with 50 indicating the most severe clinical findings related to MG) at baseline compared to end of study) at baseline compared to end of study
Myasthenia gravis Quality of Life 15 Score Efficacy Outcome | 6 months
  Change in the 15-Item Myasthenia Gravis Quality of Life Score (score 0-45, with 45 indicating the most severe clinical findings related to MG) at baseline compared to end of study) at baseline compared to end of study
Parallel Arm Comparison | 6 months
  All the above outcomes including the myasthenia gravis impairment index, quantitative myasthenia gravis score, myasthenia gravis activities of daily living, myasthenia gravis composite score, myasthenia gravis quality of life 15 score in patients receiving de novo administration starting SCIG directly with those starting with a loading dose of IVIG followed by SCIG administration will be compared.
Safety and Tolerability: total number of adverse events | 6 months
  o evaluate the adverse event profile of high dose (20% Cuvitru) SCIG in MG and compare this with existing published adverse events of 20% high-dose SCIG in neuromuscular diseases. Specifically the total number of adverse events as defined in Part C, Division 5 of the Health Canada Food and Drug Regulations will be compared to existing published adverse events of 20% SCIG and the total number of adverse events occuring in the IVIG vs SCIG arms will also be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Katzberg, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada